CLINICAL TRIAL: NCT06854146
Title: Study on the Development and Prognosis of Gastric Cancer Based on Environmental Factors and Macrogenome
Brief Title: The Effect of Environmental Factors on Gastric Cancer Based on Macrogenome
Status: Active, not recruiting | Type: Observational
Sponsor: Dong Peng (Other)
Responsible Party: Sponsor-Investigator, Dong Peng, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2024-444-01
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancers; Air Pollution
Keywords: Gastric Cancer; Macrogenome; Environmental Pollution; Air Pollution
MeSH Terms: conditions — Stomach Neoplasms | interventions — Diet, Healthy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — stool and serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- gastric cancer group: patients diagnosed with gastric cancer
  Interventions: Diagnostic Test: gastric cancer
- control group: healthy participants
  Interventions: Diagnostic Test: healthy

INTERVENTIONS:
Diagnostic Test: gastric cancer — patients diagnosed with gastric cancer
  Groups: gastric cancer group
Diagnostic Test: healthy — healthy participants
  Groups: control group

SUMMARY:
The objectives of this study were to clarify how environmental factors such as air pollution affect the occurrence and development of gastric cancer; to identify patient-specific macrogenomic markers of gastric cancer; and to investigate the mechanism of gastric cancer development based on environmental factors and macrogenomic data.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* patients with preoperative diagnosis of gastric cancer confirmed by pathologic biopsy;
* no chemotherapy, radiotherapy, targeted and immunotherapy, etc. before enrollment;
* willing to participate in the study and sign the informed consent form;
* complete clinical data.

Exclusion Criteria:

* concurrent primary malignant tumor other than gastric cancer;
* patients with systemic diseases, such as severe cardiopulmonary;
* insufficiency, that affect the choice of treatment plan;
* not suitable for enrollment as assessed by the investigator;
* incomplete clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with preoperative diagnosis of gastric cancer confirmed by pathologic biopsy and 1:1 participants with no history of malignancy were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From date of diagnosis until the date of death from any cause or or loss to follow-up, whichever came first, assessed up to 60 months
  Description: Time from diagnosis to death from any cause, measured via medical records and follow-up interviews.
  Unit: Months

SECONDARY OUTCOMES:
Gut microbiome composition differences assessed by shotgun metagenomic sequencing | Tissue samples collected intraoperatively, sequencing completed within 1 week post-surgery.
  Measuring Tool: Shotgun metagenomic sequencing (Illumina NovaSeq 6000). Analysis Parameters: Alpha diversity (Shannon index); Beta diversity (Bray-Curtis dissimilarity); Differential abundance of bacterial species (ANCOM-BC).
  Unit: Relative abundance (%) / Diversity indices.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data sharing is not permitted by the Ethics Committee of the First Affiliated Hospital of Chongqing Medical University.